CLINICAL TRIAL: NCT02988778
Title: Phase III, Multicenter, Randomized, Simple-blinded, Parallel Groups to Evaluate Non Inferiority of Noex® 50µg Versus Busonid® 50µg in Treatment of Allergic Persistent Rhinitis Moderate to Severe
Brief Title: Clinical Study, Non Inferiority Between Noex® 50µg Versus Busonid® 50µg in Treatment of Allergic Rhinitis
Acronym: RINEX50
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: regulatory strategy
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EF149
Record Dates: First submitted 2016-11-28; First posted 2016-12-09 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2017-08

CONDITIONS: Rhinitis, Allergic, Perennial
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonid 50mcg (Noex) (Experimental): Budesonid 50mcg (Noex), 2 atomizations in each nostril by the morning and during the night, total of 400 mcg per day.
  Treatment of 28 days.
  Interventions: Drug: Budesonid 50mcg (Noex)
- Budesonid 50mcg (Busonid) (Active Comparator): Budesonid 50mcg (Busonid), 2 atomizations in each nostril by the morning and during the night, total of 400 mcg per day.
  Treatment of 28 days.
  Interventions: Drug: Budesonid 50mcg (Busonid)

INTERVENTIONS:
Drug: Budesonid 50mcg (Noex) — Suspention to nasal use, 2 atomization in each nostril during the morning and at night.
  Arms: Budesonid 50mcg (Noex)
Drug: Budesonid 50mcg (Busonid) — Suspention to nasal use, 2 atomization in each nostril during the morning and at night.
  Arms: Budesonid 50mcg (Busonid)

SUMMARY:
This study is to evaluate non inferiority of Eurofarma budesonide nasal spray x referral Astrazeneca budesonide. Half patients will receive Eurofarma medication and half patients will receive Astrazeneca medication. There is no placebo group.

DETAILED DESCRIPTION:
Budesonide is a medicine already very used and registered about 20 years. Eurofarma has the intention to collect more data about safety and efficacy and present them to local authority.

This study was draw to treat patients with persistent rhinitis moderate to severe in sites located locally in Brazil.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12
2. History of allergic persistent rhinitis moderate to severe at least 2 years
3. Proved allergic using PRICK or RAST test
4. Nasal symptoms (NIS) > 3 and nasal obstruction >1
5. Indication of nasal corticosteroids use
6. Washout of nasal corticosteroids for 14 days
7. ICF

Exclusion Criteria:

1. Other types of rhinitis
2. Asthma non controlled
3. Use of oral/injectable corticoids 30 days before screening
4. patients not eligible to complete diaries
5. patients with allergy to any substance of medicines
6. non controlled disease

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Demonstrate non inferiority of Noex using the questionnaire Nasal Index Score (NIS) | 28 days
  Using the questionnaire Nasal Index Score (NIS)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Acir Crippa Junior, MD, Principal Investigator — Allergisa Pesquisa Dermato-Cosmetica LTDA
Locations (1):
- Alexandra Dumont, Campinas, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Undecided, but could be shared upon investigator's request